CLINICAL TRIAL: NCT06347354
Title: Permanence of Indocyanine Green in Axillary Lymph Nodes 3 Weeks After Subdermal Injection in Patients With Braast Cancer and Metastatic Lymph Nodes (FLUO)
Brief Title: Permanence of Indocyanine Green in Axillary Lymph Nodes 3 Weeks After Subdermal Injection in Patients With Breast Cancer and Metastatic Lymph Nodes
Acronym: FLUO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRO-2024-15
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subdermal injection of 2,5 mg (1 cc) of ICG (Experimental): Subdermal injection of 2,5 mg (1 cc) of ICG will be performed 3 weeks before surgery
  Interventions: Drug: Indocyanine green

INTERVENTIONS:
Drug: Indocyanine green — Subdermal injection of 2,5 mg (1 cc) of ICG

SUMMARY:
In the case of a pre-operative diagnosis of ductal carcinoma in situ (DCIS), sentinel lymph node biopsy is generally not indicated whereas it is considered standard clinical practice for patients with clinical stage I-II infiltrating breast cancer who have clinically negative axillary lymph nodes or clinically suspicious lymph nodes with negative needle aspiration findings. It is not uncommon that, in patients with ductal carcinoma in situ at preoperative diagnosis, there may be an upgrade on definitive histological examination due to the identification of foci of infiltration (about one-fifth of cases), requiring axillary lymph node biopsy in a second surgery. Prospective studies have shown that the sentinel lymph node identification rate after recent breast-conserving surgery is suboptimal. With regard to the false negative rate (FNR), several studies demonstrated that it could be associated with different techniques used for lymph node identification. Lymph node biopsy by Indocyanine green (ICG) is capable of identifying the sentinel lymph node, however, there are no data in literature on the permanence of ICG in the lymph node system. The knowledge of this data would allow the application of this method, already considered safe for the identification of the sentinel lymph node at the time of breast surgery, also in those situations in which the sentinel lymph node biopsy is postponed due to the upgrade of definitive histological diagnosis from carcinoma in situ to infiltrating/micro-infiltrating carcinoma.The main objective of this trial is to evaluate the permanence of fluorescence at the level of axillary lymph nodes 3 weeks after subcutaneous injection in patients who are candidates to radical axillary surgery. Marking the sentinel lymph node before breast surgery in cases of DCIS with risk factors could reduce the false negative rate, allowing to increase the accuracy of the procedure in identifying the lymph node potentially involved by metastatic infiltration. In addition, the identification of the sentinel lymph node in patients who are candidates to radical axillary surgery, could increase the sensitivity of the surgery in staging axillary disease and could make the lymph node exeresis more targeted, reducing the morbidity of the surgery resulting in a better outcome for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented before starting protocol-specific procedures and follow-up, according to local regulatory requirements.
* >18 years old
* Breast cancer patients with cyto-histologically ascertained lymph node metastases and candidates for quadrantectomy/mastectomy combined with radical axillary surgery

Exclusion Criteria:

* patients allergic to Iodine or Indocyanine Green
* patients with thyroid diseases (hyperthyroidism, autoimmune thyroid adenomas)
* patients who are not candidates for radical axillary surgery
* pregnant patients
* underage patients
* interdicted patients or patients requiring a support administrator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Permanence of fluorescence at the level of axillary lymph nodes at 2-3 weeks after subcutaneous injection of Indocyanine Green (2.5 mg), in patients who will undergo radical axillary surgery | up to 3 weeks
  Frequency of patient with at least 3 fluorescent lymph nodes

SECONDARY OUTCOMES:
Identification of the total number of fluorescent lymph nodes | up to 3 weeks
  Absolute frequency of total number of fluorescent lymph nodes per patient
Differences in the qualitative assessment (intensity) of fluorescence between the removed lymph nodes: lymph nodes will be divided into group A "intense fluorescence" and group B "mild fluorescence" | up to 3 weeks
  Absolute frequency of lymph nodes in group A and in group B
Association between histological positivity for metastases in sentinel and non-sentinel lymph nodes | up to 3 weeks
  Frequency of lymph nodes with metastases resulting fluorescent
Association between the patient's demographic/clinical variables and the presence or absence of fluorescent lymph nodes | up to 3 weeks
  Frequency of fluorescent and non-fluorescent lymph nodes between subgroups of patients with different demographic and clinical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Fracon, MD, Principal Investigator — Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy